CLINICAL TRIAL: NCT07285590
Title: International Multicentric Phase II Trial to Evaluate the Efficacy and Safety of Pirtobrutinib in Combination With Rituximab in Patients With Indolent Clinical Forms of Mantle Cell Lymphoma
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Pirtobrutinib With Rituximab in Patients With Mantle Cell Lymphoma
Acronym: IMCL-2023
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Evidenze Health España (CRO) (Unknown); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMCL-2023; 2024-511983-97-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-25; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: lymphoma; Geltamo; Rituximab; Pirtobrutinib; Mantle cell lymphoma; MCL
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — pirtobrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib with rituximab (Experimental): Patients will receive a P-R combination for at least 24 cycles (C24). The first cycle of P-R will be administered at day 1 (baseline) . Pirtobrutinib discontinuation will be decided after C24, according to the MRD response and the TP53 mutational status. Rituximab treatment will end up at C23.
  Interventions: Drug: Pirtobrutinib and rituximab

INTERVENTIONS:
Drug: Pirtobrutinib and rituximab — Patients will receive the study treatment (P-R combination) at day 1 (baseline) and during the treatment period (C24). Pirtobrutinib discontinuation per protocol will be decided after C24, according to the MRD response and the TP53 mutational status. Rituximab treatment will end up at C23.

SUMMARY:
This is a multicenter, international, open-label, single-arm phase II clinical trial designed to evaluate the activity and safety of a combination therapy with pirtobrutinib and rituximab (P-R) in treatment-naïve adult patients diagnosed with indolent clinical forms of Mantle Cell Lymphoma (MCL). The study applies a Simon's two-stage design, with an interim analysis after the first 16 patients to determine continuation based on complete remission rate (CRR) after 6 cycles.

DETAILED DESCRIPTION:
The current evidence obtained from clinical trials exploring the incorporation of BTK inhibitors in first-line treatment of MCL points toward a clear significant improvement in both patient responses and progression-free survival. Until new data from randomized clinical trials become available, the inclusion of new combinations of BTK inhibitors with chemoimmunotherapy or with new targeted combinations alone, remains a matter of debate. In addition, there is some concern regarding the additional toxicity associated with some of these combinations, which could be ameliorated by a fixed duration of treatment or by the use of newer generation BTK inhibitors, associated with significantly better tolerability. The new non-covalent BTK inhibitor pirtobrutinib has recently shown more promising activity in MCL relapsed/refractory to prior covalent BTK inhibitors therapy, and also with very favourable safety profile (3% of discontinuations due to drug-induced adverse events). Pirtobrutinib could be a very interesting drug to be tested in the upfront setting to try to sort out the significant toxicity more frequently observed with covalent BTK inhibitors. Indeed, indolent clinical forms of MCL that represent around 20% of new MCL diagnosis could be particularly suitable to receive pirtobrutinib as a first-line treatment in combination with rituximab in order to maximize responses and the rate of undetectable molecular minimal residual disease while improving the treatment tolerance. This combination could also limit treatment duration, except for MRD detectable and TP53 mutated cases, according to the data shown in the IMCL-2015 trial. By testing pirtobrutinib in combination with rituximab in a population of indolent MCL patients, the investigators aim to improve and refine the potential new standard treatment for this particular subset of MCL patients. Moreover, the Sponsor plan to conduct a clinical study that will allow not only a deep molecular MRD analysis but also a thorough biological study with different bulk and single-cell level multi-omic platforms in order to gain insight into pirtobrutinib performance in indolent clinical forms of MCL. For this purpose, the Sponsor have designed a multicenter, international, open-label, phase II clinical to assess the efficacy of pirtobrutinib in combination with rituximab in patients with indolent MCL.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years of age).
2. Written informed consent must be obtained before any study-specific assessment is performed.
3. Subjects with confirmed diagnosis of Mantle Cell Lymphoma according to the International Consensus Classification, (ICC) 2022] or World Health Organization (WHO) Classification 2022. Classical, small-cell variants and marginal-zone variants can be included.
4. Naïve patients for MCL management (no prior therapies, excluding diagnostic splenectomy)
5. Asymptomatic patients
6. Eastern Cooperative Oncology Group (ECOG) performance status <2 (0-1)
7. Clinical stage I-IV according to the Ann Arbor classification with no symptoms attributable to MCL
8. Patients with a leukemic non-nodal presentation with mainly bone marrow or peripheral blood involvement are eligible. Other asymptomatic clinical presentations are acceptable in case of low tumour burden, including MCL with lymph node enlargement ≤ 3 cm in the largest diameter and with low proliferation index (Ki67 < 30%)
9. The following laboratory values at screening:

   * Neutrophil count ≥ 1×109/L, Haemoglobin level ≥ 100 g/L and platelet count ≥100×109/L
   * Transaminases (AST and ALT) ≤ 3 x ULN
   * Total bilirubin ≤1.5 x ULN unless bilirubin rise is due to Gilbert's disease
   * Calculated creatinine clearance ≥ 30 ml/min according to Cockcroft/Gault Formula (140 - age) × body weight (kg) × 0.85 (if female)/ serum creatinine (mg/dL) × 72
   * Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) and prothrombin (PT) or (international normalized ratio (INR) not greater than 1.5 x ULN.
10. Stable disease without evidence of clinical progression for at least 3 months. Patients in prolonged observation may be included (over 3 months).
11. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use highly effective contraception from the start of study treatment (See Appendix 4), during the treatment period and for at least 1 month following the last dose of pirtobrutinib and for 12 months following treatment with Rituximab.
12. Male patients must use highly effective contraception (if sexually active with a female of child-bearing potential) according to the recommendations provided by the Clinical Trial Facilitation and Coordination Group (CTFG), from start of study treatment, during the treatment period, and for at least 1 month following the last dose of pirtobrutinib and for 12 months following treatment with rituximab.
13. Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
14. Not included in other clinical trial or treated with an experimental drug unrelated to MCL within the past 2 years

Exclusion Criteria:

1. Subjects with aggressive histological variants: blastoid and pleomorphic variants of MCL
2. B-cell monoclonal lymphocytosis with MCL phenotype
3. Presence of B symptoms or any relevant symptoms related to the MCL.
4. Nodal clinical forms with lymph node enlargement > 3 cm (largest diameter).
5. Organ dysfunction related to MCL including creatinine level > 2 mg/dl or altered liver biochemistry (> 3x ULN).
6. Serum LDH over ULN
7. Known central nervous system (CNS) infiltration.
8. Expected MCL therapy requirement in a short time (< 3 months)
9. Anticoagulation requirement with vitamin K antagonists
10. History of bleeding diathesis
11. Past medical history of stroke or intracranial haemorrhage within 6 months prior to inclusion.
12. Significant cardiovascular disease defined as: i) unstable angina or acute coronary syndrome within the past 2 months prior to randomization; ii) history of myocardial infarction within 3 months prior to randomization or documented LVEF by any method of ≤ 40% in the 12 months prior to inclusion; iii) ≥ Grade 3 NYHA functional classification system of heart failure; iv) Uncontrolled or symptomatic arrhythmias.
13. Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33). Correction of suspected drug-induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation. Correction for underlying bundle branch block (BBB) allowed.

    NOTE: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
14. Patients who have tested positive for Human Immunodeficiency Virus (HIV) are excluded due to risk of opportunistic infections with both HIV and BTK inhibitors. For patients with unknown HIV status, HIV testing will be performed at Screening and result must be negative for enrolment.
15. Known active hepatitis B virus (HBV) infection based on criteria below: Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require a negative hepatitis B polymerase chain reaction (PCR) evaluation before inclusion. Patients who are HBV DNA PCR positive will be excluded. Prophylactic antiviral treatment will be required in the patients with positive anti-HBc finally eligible.
16. Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before inclusion. Patients who are hepatitis C RNA positive will be excluded.
17. Known active cytomegalovirus (CMV) infection. Unknown or negative status are eligible.
18. Concomitant or previous malignancies the last 2 years other than basal skin cancer or in situ uterine cervix cancer.
19. Major surgery within 4 weeks of inclusion.
20. Vaccinated with live, attenuated vaccines within 4 weeks of inclusion.
21. Active uncontrolled auto-immune cytopenia (e.g., autoimmune haemolytic anaemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrolment to maintain adequate blood counts.
22. Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or any other clinically significant active disease process which in the opinion of the investigator may pose a risk for patient participation (screening for chronic conditions is not required).
23. Known hypersensitivity to any of the excipients of Pirtobrutinib or Rituximab or any intended study medications.
24. Females who are pregnant or breastfeeding or plan to become pregnant or initiate breastfeeding during the study or within 1 month of the last dose of pirtobrutinib or 12 months of the last dose of rituximab.
25. Patients unable to take oral medication or with clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Pirtobrutinib in combination with rituximab after 6 cycles | At the end of Cycle 6 (each cycle is 28 days)
  To assess the activity of Pirtobrutinib in combination with rituximab (P-R) as a therapeutic alternative to immunochemotherapy (R-Bendamustine or R-CHOP regimen) in patients with an indolent clinical presentation of MCL. The primary objective will be assessed by the complete remission rate (CRR), defined as the percentage of patients who achieve a complete response (CR) at the end of Cycle 6 of the P-R combination according to the Lugano Classification.

SECONDARY OUTCOMES:
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of ORR | At month 6, month 12 and month 24.
  The activity of P-R combination will be assessed in the overall population according to the Lugano Classification in terms of:
  • overall response rate (ORR), defined as the percentage of patients who achieved partial response (PR) or complete response (CR) according to the Lugano Classification criteria.
Evaluation of MRD | After cycle 6, cycle 12, cycle 30, cycle 36, cycle 42, cycle 48 (each cycle is 28 days), and End of treatment (28 days after las administration of Study drug).
  To evaluate and compare the MRD detection ability of different MRD assays. The sensitivity, specificity, false positive and negative rates of MRD assays: Allele-specific oligonucleotide real-time quantitative Polymerase chain reaction (ASO-qPCR) and New Generation Sequencing (NGS) based assays.
To determine the safety and tolerability of P-R combination | Baseline, during all the cycles day 1 visit (each cycle is 28 days) and at EoT (28 days afert las administration of Study drug).
  The safety of P-R combination will be assessed by terms of Adverse Events (AEs), Severe Adverse Events (SAEs), Suspected Unexpected Adverse Reactions (SUSARs) during the P-R treatment, and second neoplasms and other serious events G≥3 occurring after treatment discontinuation. All AEs will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
To assess the patient Health-related Quality of Life (HRQoL) | Between baseline and month 6, month 12, and month 24 and End of Study (month 48)
  This objective will be evaluated descriptively. The changes in the total score in patient HRQoL measured by patient reported outcomes (PRO):
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core (EORT-QLQ-C30): This questionnaire is a self-administered tool specifically developed to assess the quality of life in treated cancer patients participating in international clinical trials. It is composed of both multi-item scales and single-item measures. It consists of 30 items grouped into three multi-items measures: i) functional scales (items 1-7, 20-27), ii) symptom scales (items 8-19, 28), and (3) global health status (items 29 and 30). Items from 1 to 27 are ranked from 1 (not at all) to 4 (very much). Items 29 and 30 are ranked from 1 (very poor) to 7 (excellent). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
To assess the patient Health-related Quality of Life (HRQoL). | Between baseline and month 6, month 12, and month 24 and End of Study (month 48)
  This objective will be evaluated descriptively. The changes in the total score in patient HRQoL measured by patient reported outcomes (PRO):
  The Functional Assessment of Cancer Therapy-Lymphoma (FACT)-Lym questionnaire (version 4): This questionnaire is a self-administered tool that specifically evaluates the Lymphoma therapy in adult patients. It consists of 42 5-points Likert-type items, ranked from 0 (not at all) to 4 (very much).
To perform a comprehensive biological characterization of cases with an indolent clinical presentation of MCL | After cycle 6, cycle 12, cycle 18, cycle 24, cycle 30, cycle 36, cycle 42 and cycle 48 (Each cycle is 28 days)
  Longitudinal characterization of tumor samples prior onset of Pirtobrutinib-Rituximab and at relapse or progression (peripheral blood, plasma, bone marrow and lymph node or other tissues involved) in addition to sequential follow-up (peripheral blood and plasma samples). The biological characterization will include bulk and single-cell level multi-omic techniques.
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of CRR | At months 12 and 24
  The activity of P-R combination will be assessed in the overall population according to the Lugano Classification in terms of:
  • Complete response rate (CRR) at 12 and 24 months in overall population.
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of MRD response | At the end of Cycle 6, Cycle 12 and Cycle 24 (each cycle is 28 days)
  The rate of undetectable MRD, defined as the percentage of patients with undetectable MRD, by Allele-specific oligonucleotide real-time quantitative Polymerase chain reaction (ASO-qPCR) and New Generation Sequencing (NGS) based assays according to the response assessment (Lugano Classification criteria) after Cycle 6, Cycle 12 and Cycle 24.
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of MRD response: | At the end of Cycle 6, Cycle 12 and Cycle 24 (each cycle is 28 days)
  The time to achieve an undetectable MRD and the median duration of the undetectable MRD response in P-R responding patients.
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of clinical and molecular response duration and survival. | From the start of the study treatment with P-R until the date of first documented progression, recurrence or death, whichever came first, assessed up to 48 months
  Time-to-event variables, (calculated in the overall population):
  Duration of response (DoR), defined as the time from the documentation of tumor response to disease progression or death, in the event of no documented recurrence, or start of a new anti - lymphoma treatment because of refractory or persistent disease.
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of clinical and molecular response duration and survival. | From the start of the study treatment with P-R until the date of first documented progression, recurrence or death, whichever came first, assessed up to 48 months
  Time-to-event variables, (calculated in the overall population):
  Progression-free survival (PFS), defined as the time between start of study treatment with P-R and the first documentation of recurrence, progression, or death in the event of no documented recurrence, or start of a new anti - lymphoma treatment, due a refractory or persistent disease.
To evaluate the activity of Pirtobrutinib-Rituximab combination along time in terms of clinical and molecular response duration and survival. | From the start of the study treatment with P-R until the date of death
  Time-to-event variables, (calculated in the overall population):
  Overall survival (OS), defined as the time between the start of treatment and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Giné Soca, Principal Investigator — Hospital Clinic of Barcelona
Locations (16):
- Portugal (2):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Lisbon District
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon, Lisbon District
- Spain (14):
  - INSTITUT CATALÀ D'ONCOLOGIA (ICO). Hospital Germans Trias I Pujol., Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Institut Català d'oncologia de L'Hospitalet (ICO-L'Hospitalet), L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Clínica Universidad Navarra, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Clínica Universidad Navarra, Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in hematology diseases. All individual data collected during the trial will be available. Data shared will be coded, with no PHI included. Study protocol, statistical analysis plan, informed consent form and clinical study report will be also available. Information will be available beginning 6 months after final publication with no end date established. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting 6 months after article publication. Access to trial IPD can be requested by qualified researchers and will be provided following review and approval of a research and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact to GELTAMO though the web page: https://www.geltamo.com/contacto
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Information will be available beginning 6 months after final publication with no end date established
Access Criteria: Access to trial IPD can be requested by qualified researchers and will be provided following review and approval of a research and execution of a Data Sharing Agreement (DSA).
URL: https://www.geltamo.com/contacto

REFERENCES:
- See also: Geltamo Web page — https://www.geltamo.com/